CLINICAL TRIAL: NCT02528669
Title: Measuring Patient Ambulation in Post-Operative Recovery
Brief Title: Patient Ambulation in Post-Op Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Savvysherpa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1024875
Record Dates: First submitted 2015-07-31; First posted 2015-08-19 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2015-05

CONDITIONS: Physical Activity
Keywords: accelerometer; patient ambulation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RX Navigait (Experimental): Individuals in this group will be given an activity tracking device that receives and displays walking reminders and daily walking goals. In addition, they will be given additional education about the benefits of walking. The device will track daily steps taken, minutes of walking, and frequency of walking bouts throughout the day.
  Interventions: Device: RX Navigait
- Control Group (No Intervention): Participants in this group will be given an activity tracking device that receives and displays walking reminders and daily walking goals but will not receive additional education regarding the benefits of walking. The device will track daily steps taken, minutes of walking, and frequency of walking bouts throughout the day.

INTERVENTIONS:
Device: RX Navigait — The RX Navigait is an accelerometer that tracks the number to steps taken, duration of walking, and time of walking. In addition, this device sends messages to patients regarding daily walking goals and walking reminders.
  Arms: RX Navigait

SUMMARY:
The purpose of this study is to create a platform that accurately measures and reports patient physical activity before a procedure, during the hospital stay, and after discharge from the hospital.

DETAILED DESCRIPTION:
Early ambulation in post-operative patients has shown benefits including shorter length of stay and/or fewer complications. Accelerometers have been found as useful instruments in encouraging ambulation in patients. Accelerometers are non-invasive devices that can evaluate changes in movement, gait, and ambulatory activity. Although these devices can be beneficial, little research exists on the best way to engage patients in ambulation, how to develop a standard ambulation protocol, and the best algorithms to measure ambulation post-operation. This study seeks to develop a standardized activity tracker and program that will encourage patient ambulation and allow patients and healthcare providers to view the progress of daily walking goals.

A total of 3,000 patients will be asked if they would like to participate in this study. A healthcare provider will explain to the patient the benefits of getting out of bed, sitting, and walking after an invasive procedure. Patients who decide to participate will be given an accelerometer during their pre-operation visit or after their surgery while still in the hospital. Patients will be asked to wear the accelerometer continuously during waking hours. The accelerometer will provide patients with daily walking goals, reminders of when it is time to walk, track step count, record time of walk, and duration of walk. Patients will be asked to wear the accelerometer until their post-op visit (about 30 days).

The following data points will be analyzed:

* Relationship between ambulation and patient outcomes
* Relationship between ambulation and other health factors
* Effectiveness of prototype platform to motivate and monitor patient activity

ELIGIBILITY:
Inclusion Criteria:

* Patients of physician study investigators

Exclusion Criteria:

* Patients whose physicians find they are unfit to participate in a walking program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2016-10-10 (Actual); Study Completion 2016-10-10 (Actual)

PRIMARY OUTCOMES:
Patient Ambulation (number of steps, frequency, time) | Up to 3 months

SECONDARY OUTCOMES:
Accuracy of accelerometer algorithms measuring post operation walking | Up to three years
Number of patients completing ambulation program | Up to three years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ott, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States